CLINICAL TRIAL: NCT00166543
Title: A Phase II, Randomized, Double-Blinded Efficacy and Safety Study of Three Doses of TAS-108 Administered Orally in Postmenopausal Patients With Locally Advanced or Locally Recurrent Inoperable or Progressive Metastatic Breast Cancer Following Standard First-Line Endocrine Therapy
Brief Title: Three Doses of TAS-108 to Treat Recurrent or Recurrent Inoperable Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SRI International (Industry)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2216-03; TAS108-0004; NCT00687557 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: locally advanced breast carcinoma; locally recurrent inoperable breast carcinoma; progressive metastatic breast carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — TS 108

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- TAS-108 40 mg (Experimental)
  Interventions: Drug: TAS-108
- TAS-108 80 mg (Experimental)
  Interventions: Drug: TAS-108
- TAS-108 120 mg (Experimental)
  Interventions: Drug: TAS-108

INTERVENTIONS:
Drug: TAS-108

SUMMARY:
This study is being done to find out how safe TAS-108 is and how well TAS-108 works on recurrent or recurrent inoperable breast cancer.

DETAILED DESCRIPTION:
The objective of this study is to investigate the efficacy and safety of TAS-108 administered in postmenopausal patients with locally advanced or locally recurrent inoperable or progressive metastatic breast carcinoma who have previously responded to one or two standard endocrine therapies, with or without one prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females
* Histologically or cytologically confirmed diagnosis of breast carcinoma
* Locally advanced or locally recurrent inoperable or metastatic breast carcinoma with documented disease progression
* Has laboratory documentation of positive estrogen receptor (ER) and/or progesterone receptor (PgR) status, and has responded to the standard first or second line hormonal anti-tumor therapy given
* Has received and whose disease progressed after one or two prior systemic hormonal anti-tumor therapies
* Performance status of greater than or equal to 2 on the Zubrod scale
* Predicted life expectancy of greater than or equal to 12 weeks
* Must give written informed consent
* Measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Absolute granulocyte count of greater than 1,500/meqL, platelet count greater than 75,000/meqL, and a hemoglobin of greater than 10 g/dL
* Adequate liver and renal function as defined by a bilirubin of less than 1.5 times the upper limit of normal and a creatinine of less than 1.5 times the upper limit of normal
* Transaminases must be less than 2.5 times the upper limit of normal except for patients with liver metastases who may have transaminases less than 5 times the upper limit of normal.
* The patient has recovered from all previous anti-cancer treatment related to toxicities to at least Grade 1.
* All previous investigational drugs must be stopped at least four weeks before commencement of treatment with TAS-108.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2004-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of TAS-108 administered on this schedule | Up to 4 years and 3 months
  Treatment-emergent adverse events, serious adverse events, bone mineral density
To investigate the comparative concentrations of TAS-108 and its metabolites in tumor tissue and blood at steady-state | Up to 4 years and 3 months
To determine the time to progression of TAS-108 administered on this schedule | Up to 4 years and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James N. Ingle, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States